CLINICAL TRIAL: NCT06925308
Title: Course of Face-to-face Interactions in Adults With Autism: An Exploratory Mixed Methods Experimental Design
Brief Title: Course of Face-to-face Interactions in Adults With Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dimence Groep (Unknown)
Responsible Party: Principal Investigator, Jos Boer, MSc, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 559902
Record Dates: First submitted 2025-03-28; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder (ASD); Neurotypical
Keywords: Eye contact; Autism Spectrum Disorder; ASD; Experiment; Neurotypical; Interaction; Physiology; Reflection
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Social interaction (Experimental): Received intervention is a social interaction on which is reflected afterwards, in adults with and without autism, living in The Netherlands.
  Interventions: Behavioral: Conversation

INTERVENTIONS:
Behavioral: Conversation — The design consists of two parts. In the first part, the researcher will have a conversation (with a formal and informal phase, where the subject will be given the idea that only the formal part is part of the study) with an adult with ASD during which covert recordings of the subject's eye behavior will be made, and in addition skin conductance and duration/frequency of eye contact of the subject will be recorded, without the subject knowing that this is intended for the purpose of studying eye contact. In the second part, the researcher and subject will watch the covert recording of the subject's eye behavior, during which the subject's skin conductance will be recorded and details of the subject's behavior as seen by the researcher.

SUMMARY:
This research explores how adults with autism make eye contact during formal and informal interactions; to what extent the nature of a conversation influences how eye contact is made in terms of length, frequency and overall presentation. Also what physiological responses to eye contact are, in order to determine to what extent eye contact leads to an increased, decreased or unchanged stress level. In addition, to gain insight into the similarities and differences in how people with ASD respond to eye contact of others compared to their own eye contact.

DETAILED DESCRIPTION:
This research explores how adults with autism make eye contact during formal and informal interactions; to what extent the nature of a conversation influences how eye contact is made in terms of length, frequency and overall presentation. Also what physiological responses to eye contact are, in order to determine to what extent eye contact leads to an increased, decreased or unchanged stress level. In addition, to gain insight into the similarities and differences in how people with ASD respond to eye contact of others compared to their own eye contact.

The research design chosen is an exploratory mixed methods study, which was developed in co-design with an expert by experience. The design consists of two parts. In the first part, the researcher will have a conversation (with a formal and informal phase, in which the subject will be given the idea that only the formal part is part of the research) with an adult with ASD, during which hidden recordings of the subject's eye behavior will be made, and in addition, skin conductance and duration/frequency of the subject's eye contact will be recorded, without the subject knowing that this is intended for research into eye contact. In the second part, the researcher and subject watch the hidden recording of the subject's eye behavior, during which the subject's skin conductance will be recorded and special features of the subject, as seen by the researcher. Both the arrangement of the subjects and researcher, as well as the physiological measurements, will be tested in advance.

ELIGIBILITY:
Inclusion criteria

* Neurotypical adults and adults with an ASD, determined according to an internationally recognized classification system.
* Able to understand the instructions.
* Motivation to participate in research.

Exclusion criteria

* No good command of the Dutch language.
* Use of alcohol and/or recreational drugs during the research.
* Mentally too unstable to participate in the research.
* Familiarity with treatment in the VGZ.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of eye contact in adults with autism, measured with video, audio and push button. | Baseline
  The research consists of two parts. During the first part, the conversation, the frequency of eye contact will be investigated. This will be measured by video recordings of the eye region combined with the pressing of a push button by the researcher at moments when eye contact is present.
  Data will be analyzed using software programs Observer XT and Matlab for the integration of push button, video recordings and audio recordings.
Duration of eye contact in adults with autism, measured with video, audio and push button. | Baseline
  The research consists of two parts. During the first part, the conversation, the duration of eye contact will be investigated. This will be measured by video recordings of the eye region combined with the pressing of a push button by the researcher at moments when eye contact is present. Data will be analyzed using software programs Observer XT and Matlab for the integration of push button, video recordings and audio recordings.
Arousal during eye contact in adults with autism, measured with skin conductance | Baseline
  The research consists of two parts. During the first part, the arousal during eye contact will be investigated. This will be measured by a skin conductance meter and analysed with the software program VSRRP.
Arousal during reflection on ones own eye contact in adults with autism, measured with skin conductance | Baseline
  During the second part, the reflection on video recordings of ones own eye contact in aduls with autism, the degree of arousal to seeing their own eye contact will be investigated. For this, skin conductance meter will be used and analysed with the software program VSRRP.
Reflection on ones own eye contact in adults with autism, measured with video and audio | Baseline
  During the second part, reflection first part, it will be investigated how subjects respond with words. For this, audio and video recordings will be used. Data analysis will be conducted with use of thematic analysis and software programs Atlas.ti, Microsoft Excel and Microsoft Word.

CONTACTS AND LOCATIONS:
Overall Officials: Nynke Boonstra, Professor, Study Chair — UMC Utrecht
Locations (1):
- Dimence Groep, Deventer, Overijssel, Netherlands